CLINICAL TRIAL: NCT00399789
Title: A Phase 1/2 Trial of Perifosine in the Treatment of Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 201
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2012-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-Small-Cell Lung; Perifosine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perifosine 150 mg qd (Active Comparator): A daily dose of 150 mg to be given in one dose at bedtime. If patients experience no grade 2 toxicities during their first month of therapy, the dose will be escalated to 200 mg to be given in one dose at bedtime.
  Interventions: Drug: Perifosine
- Perifosine 900 mg per week (Active Comparator): A weekly dose of 900 mg to be divided into three doses of 300 mg each. If patients experience no grade 2 toxicities during their first month of therapy, the dose will be escalated to 1,200 mg divided into four doses of 300 mg.
  Interventions: Drug: Perifosine
- Perifosine 50 mg tid (Active Comparator): A daily dose of 150 mg to be divided into three doses of 50 mg each. If patients experience no grade 2 toxicities during their first month of therapy, the dose will be escalated to 200 mg divided into four doses of 50 mg.
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine — Perifosine will be tested in 3 dose forms

SUMMARY:
This is a study of the drug perifosine that consists of 2 parts. The first part of this study was designed to determine the highest dose of perifosine that can be administered to people every week without severe or prolonged nausea, vomiting and diarrhea. This study started with patients taking 900 mg/week and went up to 1800 mg/week. Part I of this study is completed. The MTD had been determined and incorporated in Part II.

The goals in Part II are to:

1. Compare the gastrointestinal toxicity of 3 different dose-schedules and
2. Obtain preliminary information on the response rate of perifosine in non-small cell lung cancer.

DETAILED DESCRIPTION:
The primary purpose of Part I of this study was to determine the maximum dose of perifosine that can be administered with tolerable gastrointestinal toxicity; and to obtain preliminary information on the response rate of perifosine in non-small cell lung cancer. In addition, the trial was and is designed to provide some insight into the nature of the anti-tumor effect, the time to response, and dose-schedules that should be used in future trials.

Part 2 - In the second part of this study, patients will be randomized to one of 3 dose-schedules of perifosine and to test if the response rate of perifosine in non small cell lung cancer is > 10% in any of the 3 arms of the study. The study is not designed to compare the response rates in the 3 arms of the trial, but toxicities will be compared. The regimens are:

* A weekly dose of 900 mg to be divided into three doses of 300 mg each. If patients experience no grade 2 toxicities during their first month of therapy, the dose will be escalated to 1,200 mg divided into four doses of 300 mg.
* A daily dose of 150 mg to be divided into three doses of 50 mg each. If patients experience no grade 2 toxicities during their first month of therapy, the dose will be escalated to 200 mg divided into four doses of 50 mg.
* A daily dose of 150 mg to be given in one dose at bedtime. If patients experience no grade 2 toxicities during their first month of therapy, the dose will be escalated to 200 mg to be given in one dose at bedtime.

Patients receiving weekly perifosine will receive prophylactic antiemetics. Patients receiving daily perifosine will not routinely receive prophylactic antiemetics unless they experience nausea. All patients may continue therapy unless disease progression is documented on two occasions at least 4 weeks apart. Patients who experience toxicity may continue on treatment with doses delayed or reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of non-small cell lung cancer, must have progressed despite standard therapy and must not be candidates for surgical or combined modality therapy.
* At least 18 years of age.
* Patients should have received at least one but no more than two prior chemotherapy regimens for metastatic disease. The study chairman or medical monitor will consider extenuating circumstances for patients with more than two such regimens.
* Patients must have measurable disease. Since the outcome for a patient is to be based on response using RECIST criteria, the patient must have at least one measurable lesion that can be accurately measured in at least one dimension and fit one of the following criteria: longest diameter 20 mm using conventional techniques or 10 mm with spiral CT scan.
* Patients must have a life expectancy of more than 3 months.
* Patients should have a performance status of 0 to 1 according to the ECOG criteria. However, patients with ECOG performance status of 2 may be admitted with approval from the study chairman or medical monitor.
* Female patients who are pregnant or lactating are ineligible. All females of childbearing potential must have a negative serum pregnancy test within 72 hours of treatment. Men and women of childbearing potential must agree to employ adequate contraception to prevent pregnancy while on therapy and for four weeks after the completion of treatment.
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients with rapidly progressing disease, as defined by progression within 12 weeks of initiation of the previous regimen.
* Patients receiving any other investigational agents or devices.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment) or New York Heart Assoc. class II-IV congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2004-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal toxicity of 3 different dose-schedules | 12 weeks
  The frequency of grade 2 or greater gastrointestinal toxicities between the 3 arms of the study will be observed and used to determine the best regimen

SECONDARY OUTCOMES:
Preliminary information on response rate | 3 months
  To test if the response rate of perifosine in non small cell lung cancer is > 10% in any of the 3 arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (20):
- United States (20):
  - AOI Pharmaceuticals Investigative Site, Tucson, Arizona
  - AOI Pharmaceuticals Investigative Site, Pomona, California
  - AOI Pharmaceuticals Investigative Site, Aventura, Florida
  - AOI Pharmaceuticals Investigative Site, Hollywood, Florida
  - AOI Pharmaceuticals Investigative Site, Lakeland, Florida
  - AOI Pharmaceuticals Investigative Site, Ormond Beach, Florida
  - AOI Pharmaceuticals Investigative Site, Lawrenceville, Georgia
  - AOI Pharmaceuticals Investigative Site, Galesburg, Illinois
  - AOI Pharmaceuticals Investigative Site, New Albany, Indiana
  - AOI Pharmaceuticals Investigative Site, Grand Rapids, Michigan
  - AOI Pharmaceuticals Investigative Site, Kalamazoo, Michigan
  - AOI Pharmaceuticals Investigative Site, Billings, Montana
  - AOI Pharmaceuticals Investigative Site, Albuquerque, New Mexico
  - AOI Pharmaceuticals Investigative Site, Albany, New York
  - AOI Pharmaceuticals Investigative Site, Armonk, New York
  - AOI Pharmaceuticals Investigative Site, Greenville, South Carolina
  - AOI Pharmaceuticals Investigative Site, Chattanooga, Tennessee
  - AOI Pharmaceuticals Investigative Site, Nashville, Tennessee
  - AOI Pharmaceuticals Investigative Site, Dallas, Texas
  - AOI Pharmaceuticals Investigative Site, Tyler, Texas

REFERENCES:
- [Result] Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 24, No 18S (June 20 Supplement), 2006: 13063